CLINICAL TRIAL: NCT01468688
Title: A Multi-arm Dose-finding Phase Ib Multicenter Study of Imatinib in Combination With the Oral Phosphatidyl-inositol 3-kinase (PI3-K) Inhibitor BKM120 in Patients With Gastrointestinal Stromal Tumor (GIST) Who Failed Prior Therapy With Imatinib and Sunitinib
Brief Title: A Dose-finding Study of a Combination of Imatinib and BKM120 in the Treatment of 3rd Line GIST Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571X2101; 2011-002938-39 (EudraCT Number)
Record Dates: First submitted 2011-11-06; First posted 2011-11-09 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2019-09

CONDITIONS: 3rd Line GIST
Keywords: Imatinib mesylate; BKM120; GIST
MeSH Terms: interventions — Imatinib Mesylate; NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- STI571 (imatinib mesylate) and BKM120 (Experimental): The study will comprise of 2 parts. A dose escalation and a dose expansion part. Patients will receive increasing doses of BKM120 (40, 60, 80, 100 mg) in combination with 400mg imatinib daily until maximum tolerated dose (MTD) and rapid phase 2 dose (RP2D) is determined. 35 patients will enter the expansion phase with 18 patients having a pharmacokinetic (PK) run-in period of 8 days receiving imatinib monotherapy or BKM120 monotherapy.
  Interventions: Drug: STI571
- STI571+BKM120 (Experimental): BKM120 Monotherapy 8 day run-in followed by STI571 and BKM120 combination therapy
  Interventions: Drug: STI571; Drug: BKM120
- STI571 monotherapy run-in (Experimental): STI571 Monotherapy 8 day run-in followed by STI571 and BKM120 combination therapy
  Interventions: Drug: STI571

INTERVENTIONS:
Drug: STI571
Drug: BKM120 — BKM120 combination therapy
  Arms: STI571+BKM120

SUMMARY:
The purpose of this study is to determine a maximum tolerated dose and/or recommended phase 2 dose of a combination of imatinib and BKM120 in the treatment of 3rd line GIST patients.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients ≥ 18 years of age
2. WHO performance status (PS) of 0-2
3. Histologically confirmed diagnosis of GIST that is unresectable or metastatic
4. Available tissue specimen:

   * Dose-escalation cohorts: patients must have available archival tumor tissue which can be shipped during the course of the study
   * Dose-expansion cohort: patients must have available archival tumor tissue which can be shipped during the course of the study and must agree to a fresh pre-treatment biopsy.
5. Failed prior therapy with imatinib followed by sunitinib for the treatment of unresectable or metastatic GIST. Note the following specific criteria for the two phases of the trial:

   * Dose-escalation cohorts: patients who failed prior therapy with imatinib and then have failed therapy with sunitinib. Treatment failure may be due to either disease progression on therapy (both imatinib and sunitinib) or intolerance to therapy (sunitinib). Dose-escalation cohort patients may have had additional lines of therapy not limited to imatinib and sunitinib.
   * Dose-expansion cohort: patients must have documented disease progression on both imatinib and sunitinib. In addition, patients may have had no more than two lines of prior therapy (i.e. treatment with imatinib followed by treatment with sunitinib).
   * Adjuvant imatinib will not count as a prior course of imatinib for the purposes of this criterion

Exclusion Criteria:

1. Previous treatment with PI3-K inhibitors
2. A medical history of any of the following mood disorders as judged by the Investigator or a psychiatrist:

   * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or thoughts, or homicidal thoughts (immediate risk of doing harm to others)
   * ≥ CTCAE grade 3 anxiety
3. When completing the patient questionnaires at screening:

   * Meets the cut-off score of ≥ 10 in the nine item depression scale of the Patient Health Questionnaire (PHQ-9) or a cut-off of ≥ 15 in the Generalized Anxiety Disorder Assessment (GAD 7) mood scale respectively, or
   * Selects positive response of 1, 2, 3 to question number 9 regarding potential for suicidal thoughts or ideation in the PHQ-9 (independent of the total score of the PHQ-9)
4. Severe and/or uncontrolled concurrent medical condition that, in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. acute or chronic liver, pancreatic, severe renal disease considered unrelated to study disease, chronic pulmonary disease including dyspnea at rest from any cause).
5. Poorly controlled diabetes mellitus (defined as HbA1c > 8%)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04-20 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
Frequency and characteristics of dose limiting toxicities (DLTs) at each dose level during the first cycle of therapy | 28 days (1st cycle)
  Dose limiting toxicity (DLT) will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) (v4.0.3), unless otherwise specified in the protocol.

SECONDARY OUTCOMES:
Frequency and characteristics of DLTs at each dose level during the first cycle of therapy. Type, frequency and severity of adverse drug reactions. | 28 days (1st cycle)
  Dose limiting toxicity (DLT) will be assessed using CTCAE (v4.0.3), unless otherwise specified in the protocol.
Imatinib and BKM120 plasma concentrations vs time profile, and basic PK parameters, including but not limited to AUC, Cmax, Tmax, CL/F. | 28 days (1st cycle)
Clinical benefit rate (CBR) defined as the rate of confirmed complete response (CR) or partial response (PR), or stable disease (SD) which lasts for at least 16 weeks. | 28 days (1st cycle)
  Tumor response will be determined locally by the investigator sites according to Novartis guideline on the Response Evaluation Criteria in Solid Tumors, based on RECIST Version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (2):
  - Dana Farber Cancer Institute SC (2), Boston, Massachusetts
  - Seattle Cancer Care Alliance Onc, Seattle, Washington
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Vancouver, British Columbia, Canada
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gelderblom H, Jones RL, George S, Valverde Morales C, Benson C, Jean-Yves Blay, Renouf DJ, Doi T, Le Cesne A, Leahy M, Hertle S, Aimone P, Brandt U, Schӧffski P. Imatinib in combination with phosphoinositol kinase inhibitor buparlisib in patients with gastrointestinal stromal tumour who failed prior therapy with imatinib and sunitinib: a Phase 1b, multicentre study. Br J Cancer. 2020 Apr;122(8):1158-1165. doi: 10.1038/s41416-020-0769-y. Epub 2020 Mar 9. PMID 32147671
- See also: Novartis' results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16508